CLINICAL TRIAL: NCT02735876
Title: A Randomized, Multicenter, Open Label, Phase 3 Study of Acalabrutinib (ACP-196) in Combination With Rituximab Versus Ibrutinib Versus Acalabrutinib Alone in Subjects With Relapsed or Refractory (R/R) Mantle Cell Lymphoma (MCL)
Brief Title: A Study of Acalabrutinib in Combination With Rituximab Versus Ibrutinib Versus Acalabrutinib in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-309
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: Bruton tyrosine kinase inhibitor; Btk; ACP-196; Mantle Cell Lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- acalabrutinib plus rituximab (Experimental): Acalabrutinib will be orally administered until disease progression or unacceptable toxicity. Rituximab IV infusions will be administered weekly for 4 weeks and on Day 1 of Cycle 3 through 8, and thereafter every other cycle for less than or equal to two years (approximately 200 subjects).
  Interventions: Drug: acalabrutinib; Drug: rituximab
- ibrutinib (Active Comparator): Ibrutinib will be orally administered until disease progression or unacceptable toxicity (approximately 200 subjects).
  Interventions: Drug: ibrutinib
- acalabrutinib (Experimental): Acalabrutinib will be orally administered until disease progression or unacceptable toxicity (approximately 50 subjects).
  Interventions: Drug: acalabrutinib

INTERVENTIONS:
Drug: acalabrutinib
  Arms: acalabrutinib; acalabrutinib plus rituximab
Drug: ibrutinib
  Arms: ibrutinib
Drug: rituximab
  Arms: acalabrutinib plus rituximab

SUMMARY:
This study is evaluating the efficacy of acalabrutinib in combination with rituximab (Arm 1) versus ibrutinib (Arm 2) versus acalabrutinib (Arm 3) for the treatment of relapsed or refractory (R/R) mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Pathologically confirmed mantle cell lymphoma (MCL).
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use highly effective forms of contraception during the study and for 90 days after the last dose of acalabrutinib or ibrutinib or 12 months after the last dose of rituximab (whichever is longest).
* Disease that has relapsed, or been refractory to, ≥ 1 prior treatment regimen for mantle cell lymphoma (MCL).
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

* Any history of central nervous system (CNS) lymphoma or leptomeningeal disease.
* Prior exposure to ibrutinib or to a B-cell receptor (BCR) inhibitor.
* Significant cardiovascular disease.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection.
* Known history of infection with human immunodeficiency virus (HIV).
* History of hepatitis B (HBV) infection or active infection with hepatitis C (HCV).
* Breastfeeding or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by Independent Review Committee (IRC) per the Lugano Classification for Non-Hodgkin Lymphoma (NHL). The primary analysis is a comparison of progression-free survival (PFS) between Arm 1 and Arm 2. | 48 months

SECONDARY OUTCOMES:
Investigator-assessed progression-free survival (PFS) per the Lugano Classification for Non-Hodgkin Lymphoma (NHL). | 48 months
Investigator-assessed overall response rate (ORR) per the Lugano Classification for Non-Hodgkin Lymphoma (NHL). | 48 months
Overall survival (OS). | 48 months
IRC-assessed duration of response (DOR) per the Lugano Classification for Non-Hodgkin Lymphoma (NHL). | 48 months

OTHER OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), and adverse events (AEs) leading to treatment discontinuation. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Inamdar, MBBS, Study Director — Acerta Pharma, LLC

IPD SHARING:
Plan to Share IPD: Undecided